CLINICAL TRIAL: NCT04267614
Title: Clinical Outcomes of Early Versus Delayed Management of Iraqi Patients With Rheumatoid Arthritis With Etanercept
Brief Title: This Study is to Investigate the Effect of Etanercept in Early Versus Delayed Referral for Management of Rheumatoid Arthritis Patients.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801411
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Results first posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2022-08

CONDITIONS: Arthritis Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Rheumatoid Arthritis (RA): Patients receiving etanercept from Baghdad teaching hospital registry(Rheumatology center) from 2012 till 2017. Patients were identified as receiving early versus delayed etanercept treatment.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Patients who received etanercept for RA

SUMMARY:
This study is to investigate the effect of etanercept in early versus delayed referral for management of rheumatoid arthritis patients assessing real-world patient data entered in the Iraq National Center of Rheumatology database between May 2012 and May 2017.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed RA patients.
* 18 years old and above.
* Did not receive pervious biological treatment.

Exclusion Criteria:

* Had previous biological treatment
* Use etanercept for less than 1 year

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data will be collected from the Baghdad teaching hospital registry. The Rheumatology patient registry is a prospective longitudinal multicentre cohort initiated in 2012.
Sampling Method: Non-Probability Sample
Enrollment: 1226 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of Iraq participants aged greater than or equal to (>=) 18 years, who received etanercept for at least 1 year anytime from 2012 until 2018 for treatment of rheumatoid arthritis (RA) and met American College of Rheumatology/ European League Against Rheumatism (EULAR) 2012 criteria for RA, were included in the study. Data were collected from Baghdad teaching hospital registry. Available data were evaluated in 1 month of this retrospective, observational study.
Groups:
- Etanercept: Participants with RA received etanercept for at least 1 year (anytime from 2012 until 2018) under standard real world clinical practice, were included in this study. Data for these participants were studied for 1 month in this retrospective observational study.
Period: Overall Study
Arm/Group | Etanercept
Started ((Medical records retrieved)) | 1226
Included in Analysis | 979
Completed | 979
Not Completed | 247
Not completed — Participants did not meet inclusion criteria | 132
Not completed — Lost to Follow-up | 115

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants who met the inclusion criteria to use the data for analysis for retrospective observation.
Arm/Group | Etanercept
Number analyzed (Participants) | 979
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.06 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 813
  Male | 166
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Disease Activity Score 28 (DAS28) at Month 12
Description: DAS28 was calculated from the number of swollen joints (SJC) and painful joints (PJC) using 28 joints count, the erythrocyte sedimentation rate (ESR) (in millimeters per hour [mm/hour]) and patient's global assessment (PGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated high disease activity). DAS28 less than or equal to (<=) 3.2 = low disease activity, DAS28 greater than (>) 3.2 to 5.1 = moderate to high disease activity. Participants were grouped based on early and delayed referral to management of RA with etanercept treatment. Early referral was considered when participants were referred to management of RA from 1 to 9.9 years and delayed referral was considered when participants were referred to management of RA for >9.9 years after diagnosis with RA.
Time Frame: Month 12 (from the data retrieved and observed during 1 month of this study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Etanercept: Participants With Early Referral (1 to 9.9 Year): Participants who received early etanercept treatment for RA (1 to 9.9 year after diagnosis with RA) for at least 1 year (anytime from 2012 until 2018) under standard real world clinical practice, were included in this arm. Data for these participants were studied for 1 month in this retrospective observational study.
- Etanercept: Participants With Delayed Referral (> 9.9 Years): Participants who received delayed etanercept treatment for RA (>9.9 year after diagnosis with RA) for at least 1 year (anytime from 2012 until 2018) under standard real world clinical practice, were included in this arm. Data for these participants were studied for 1 month in this retrospective observational study.
Arm/Group | Etanercept: Participants With Early Referral (1 to 9.9 Year) | Etanercept: Participants With Delayed Referral (> 9.9 Years)
Number analyzed (Participants) | 579 | 400
Units on a scale | 4.56 (1.12) | 4.9 (1.23)
Statistical Analysis 1: Comparison: Etanercept: Participants With Early Referral (1 to 9.9 Year) vs Etanercept: Participants With Delayed Referral (> 9.9 Years); Test type: Other; p < 0.05, t-test, 2 sided

2. Primary Outcome: Clinical Disease Activity Index (CDAI) Score at Month 12
Description: The CDAI is the numerical sum of 4 outcome parameters: tender joint count (TJC) and SJC based on a 28-joint assessment, PGA and physician global assessment (PhGA) assessed on 0 to 10 centimeter (cm) visual analog scale (VAS); higher scores = high disease activity. CDAI total score = 0 to 76. CDAI <= 2.8 indicates disease remission, > 2.8 to 10 = low disease activity, > 10 to 22 = moderate disease activity and > 22 = high disease activity. Participants were grouped based on early and delayed referral to management of RA with etanercept treatment. Early referral was considered when participants were referred to management of RA from 1 to 9.9 years and delayed referral was considered when participants were referred to management of RA for >9.9 years after diagnosis with RA.
Time Frame: Month 12 (from the data retrieved and observed during 1 month of this study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept: Participants With Early Referral (1 to 9.9 Year) | Etanercept: Participants With Delayed Referral (> 9.9 Years)
Number analyzed (Participants) | 579 | 400
Units on a scale | 19 (10) | 22 (11.2)
Statistical Analysis 1: Comparison: Etanercept: Participants With Early Referral (1 to 9.9 Year) vs Etanercept: Participants With Delayed Referral (> 9.9 Years); Test type: Other; p < 0.05, t-test, 2 sided

3. Other Pre Specified Outcome: Mean Change From Baseline in DAS28 at Month 12
Description: DAS28 was calculated from the SJC and PJC using 28 joints count, the ESR (in mm/hour) and PGA of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated high disease activity). DAS28 <=3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity. Participants were grouped based on early and delayed referral to management of RA with etanercept treatment. Early referral was considered when participants were referred to management of RA from 1 to 9.9 years and delayed referral was considered when participants were referred to management of RA for >9.9 years after diagnosis with RA. Baseline was defined as Day 0 before receiving etanercept.
Time Frame: Baseline, Month 12 (from the data retrieved and observed during 1 month of this study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept: Participants With Early Referral (1 to 9.9 Year) | Etanercept: Participants With Delayed Referral (> 9.9 Years)
Number analyzed (Participants) | 579 | 400
Units on a scale
  Baseline | 5.61 (1.24) | 5.79 (1.17)
  Change at Month 12 | 1.0 (1.1) | 0.9 (1.09)
Statistical Analysis 1: Comparison: Etanercept: Participants With Early Referral (1 to 9.9 Year) vs Etanercept: Participants With Delayed Referral (> 9.9 Years); Test type: Other; p < 0.05, t-test, 2 sided

4. Other Pre Specified Outcome: Mean Change From Baseline in CDAI Score at Month 12
Description: The CDAI is the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PGA and PhGA assessed on 0 to 10 cm VAS; higher scores = high disease activity. CDAI total score = 0 to 76. CDAI <= 2.8 indicates disease remission, > 2.8 to 10 = low disease activity, > 10 to 22 = moderate disease activity and > 22 = high disease activity. Participants were grouped based on early and delayed referral to management of RA with etanercept treatment. Early referral was considered when participants were referred to management of RA from 1 to 9.9 years and delayed referral was considered when participants were referred to management of RA for >9.9 years after diagnosis with RA. Baseline was defined as Day 0 before receiving etanercept.
Time Frame: Baseline, Month 12 (from the data retrieved and observed during 1 month of this study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept: Participants With Early Referral (1 to 9.9 Year) | Etanercept: Participants With Delayed Referral (> 9.9 Years)
Number analyzed (Participants) | 579 | 400
Units on a scale
  Baseline | 27.03 (11.79) | 28.55 (11.35)
  Change at Month 12 | 7.9 (6.7) | 6.5 (7.1)
Statistical Analysis 1: Comparison: Etanercept: Participants With Early Referral (1 to 9.9 Year) vs Etanercept: Participants With Delayed Referral (> 9.9 Years); Test type: Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events not collected during the study
Description: Due to non-interventional nature of study, the minimum criteria for reporting an adverse event (i.e. identifiable participant, identifiable reporter, a suspect product, and event) could not met, hence, safety data was not collected and reported.
Arm/Group | Etanercept
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT04267614/Prot_SAP_000.pdf